CLINICAL TRIAL: NCT03391921
Title: Prospective Longitudinal Study on Immunogenicity, Induction of Cellular Immune Responses and Safety of Vaccination Against HPV With the 9-valent Vaccine in HIV-positive Women (The Papillon Study)
Brief Title: Vaccination Against Human Papillomavirus (HPV) With the 9-valent Vaccine in HIV-positive Women (the Papillon Study)
Acronym: Papillon
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Saint Pierre (Other)
Responsible Party: Principal Investigator, Deborah Konopnicki, Head of clinic, Infectious Diseases Department, Centre Hospitalier Universitaire Saint Pierre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CE/17-12-06
Record Dates: First submitted 2017-12-14; First posted 2018-01-05 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: HPV - Anogenital Human Papilloma Virus Infection; HIV Infections
Keywords: vaccine; woman
MeSH Terms: conditions — HIV Infections | interventions — Vaccines

STUDY DESIGN:
Intervention Model Description: After a first open label phase evaluating tolerability of Gardasil9 in HIV-positive women and where all patients (n=50) have received three doses (0,2 and 6 months) of the 9valent vaccine against HPV from June 2018 to end of December 2018, the study will randomize participants between two between two different doses schedules: in the first schedule (ARM A), women will receive 2 doses at time 0 and 6 months and a third dose between 18-48 months if their antibody levels are insufficient; the second schedule (ARM B) will be 3 doses at 0, 2 and 6 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ARM B: 3 doses (0, 2 and 6 months) (Active Comparator): ARM B: All patients will receive the 9-valent vaccine against HPV (Gardasil9) 3 doses at 0,2 and 6 months intramuscularly
  Interventions: Biological: Vaccine
- ARM A: 2 doses (0 and 6 months ) (Experimental): ARM A: All patients will receive the 9-valent vaccine against HPV (Gardasil9) 2 doses at 0 and 6 months intramuscularly. A third facultative dose will be given if antibodies measured at month 7 are insufficent.
  Interventions: Biological: Vaccine

INTERVENTIONS:
Biological: Vaccine — All patients will receive the 9-valent vaccine against HPV (Gardasil9) intramuscularly: After a first open phase evaluating tolerability of Gardasil9, women will be randomized between two different doses schedules: in the first schedule, women will receive 2 doses at time 0 and 6 months and a third dose between 18-48 months if their antibody levels are insufficient; the second schedule will be 3 doses at 0, 2 and 6 months.

SUMMARY:
Phase IV prospective study measuring the immunogenicity (neutralizing antibody titles against each HPV vaccine genotype) of the 9-valent vaccine against HPV (Gardasil9®Merck) in HIV-positive women aged 15-40 years with fully suppressed HIV viremia on combined antiretroviral therapy.

After a first open phase evaluating tolerability of Gardasil9 (from June 2018 to December 2018), an amendment was introduced to randomize women between two different doses schedules: in the first schedule (ARM A), women will receive 2 doses at time 0 and 6 months and a third dose between 18-48 months if their antibody levels are insufficient; the second schedule (ARM B) will be 3 doses at 0, 2 and 6 months. Primary outcome is the non-inferiority of the rate of seroconversion against each HPV vaccine genotypes in women seronegative at baseline after either 2 or 3 doses of vaccination (month 7). Secondary outcomes are rate of seroconversion after 3 doses if they have received a third dose, completion of vaccine schedule, vaccine safety, antibody titles, and induction of cellular immunity against HPV contained in the vaccine, incidence of cervical HPV infection and incidence of abnormal cytology after vaccination. The safety of the vaccination (local or systemic reaction and impact on HIV viral control and immunodeficiency level) will be assessed. The cellular immune response will be assessed in a subgroup of patients.

DETAILED DESCRIPTION:
Number of patients:

Study: 200 patients: 50 in the first open label phase (june 2018 to dec 2018), then n=150 in the randomized phase starting in January 2019 Substudy on immune response analysis in a subset of patients: 40 patients and separated informed consent

Primary outcome:

Rate of seroconversion of neutralizing antibodies against each HPV vaccine genotypes namely 6/11/16/18/31/33/45/52/58 among women seronegative at baseline for HPV vaccine genotypes, by measuring neutralizing antibody against the 9 vaccine genotypes of HPV at baseline, month 7. The measure will be performed on a 10 ml tube by chemiluminescence immunoassay (cLIA) technique in Merck laboratory .Comparison of that rate at month 7 (non inferiority defined as at least 80% of seroconversion in ARM A).

Secondary outcomes:

1. Incidence of Treatment-Emergent Adverse Events (Safety and tolerability of the vaccines).

   It will be evaluated by a specific questionnaire on a phone call made by the research team to the participant and scheduled at least 48 hours and maximum 7 days after each vaccine dose; the questionnaire will evaluate whether there is any complain regarding local reaction (pain, redness, swelling, pruritus), systemic reaction (fever, malaise and fatigue) or other side effect. In case of any usual complain > mild stage, or the presence of an unusual complain, the patient will be assessed by a visit and physical examination performed by the research team. The questionnaire has been elaborated according to the published data on safety evaluation of the 9-valent vaccine.
2. The potential impact of vaccine administration on T-lymphocyte-CD4+ cell count and HIV viremia It will be assessed by measuring CD4 cell count and HIV viremia at baseline (any measure within 6 months before screening can be taken into account) and month 7. Any detectable HIVRNA >50 cp/ml will be reassessed on a second samples taken 2-4 weeks later. Any significant decrease in T-lymphocyte-CD4+ cell count (defined as a decrease by more of 5% in the percentage or >100 cells/µl) will be reassessed on a second sample taken 2-4 weeks later.
3. Measure of the geometric mean titre of specific neutralizing antibodies against each HPV vaccine genotypes (6/11/16/18/31/33/45/52/58).

   It will be assessed before vaccination, 1 month after vaccination completion (month 7) and 12 months after vaccination completion (month 18). In December 2022, the protocol was amended to add follow up at month 24,36,48 and 60.
4. The cellular immune response The cellular immune response ill be evaluated in a subset of 40 patients (aged 18-40 years old) by measuring specific T-lymphocytes-CD4+ cells expressing CD40-receptor, interleukin-2 (IL2), interferon gamma (IFN-g) or Tumor necrosis factor (TNF-alpha ) against HPV 16/18/31/52 and 58. The analysis will be performed on a peripheral blood mononuclear cell (PBMC) sample of 30 to 50 ml taken at baseline and at month 7; a separate informed consent (IC) has to be signed for this sub-analysis.
5. The incidence and prevalence rates of cervical HPV infections:

   Detection of HPV will be performed by molecular technique by the national reference center for HPV (AML, Antwerpen), performed on cervical swab taken by the gynecologist at baseline and month 18. The baseline gynecological sample might have been taken up to 6 months before the vaccination. These swabs will be sampled in all participants with previous vaginal sexually activity. In case of no previous vaginal sexual intercourse, the samples will not be taken.
6. The incidence and prevalence rates of abnormal cervical cytology:

   Cervical cytology will be performed by by the national reference center for HPV (AML, Antwerpen) on cervical swab taken by the gynecologist at baseline and month 18. The baseline gynecological sample might have been taken up to 6 months before the vaccination. These swabs will be sampled in all participants with previous vaginal sexually activity. In case of no previous vaginal sexual intercourse, the samples will not be taken.
7. Completion of vaccine schedule. Comparison of the proportion of women achieving full course of vaccine administration in each arm, namely for ARM A receiving 2 doses and for ARM B receiving 3 doses.
8. Proportion of patients needing a booster dose (i.e..a third dose) in ARM A If after 2 doses of vaccine (ARM A), the month 7 antibodies analysis shows absence of seroconversion against one of the HPV genotypes contained in the vaccine, the participant will receive a third booster dose

Number of visits:

4 to 5 mandatory visits at baseline, month 2 (not if ARM A), month 6, month 7 and month 18 plus 2 to 3 optional visits to be done in case of moderate or severe adverse reaction to vaccine administration

ELIGIBILITY:
Inclusion Criteria:

* HIV-positive woman
* Age 15-40 years
* Undetectable HIV viral load (HIVRNA <400 cp/ml) for at least 6 months (i,e: having at least two separate HIVRNA <400 cp/ml at 6 months intervals; the most recent HIVRNA <400 cp/ml may be performed with the baseline sample for the study).
* No planned pregnancy foreseen for the next 7 months and use of contraception such as condom, hormonal contraception or intrauterine device
* IC signed

Exclusion Criteria:

* Previous hysterectomy or conisation
* Previous or current biopsy-proven cervical, vulvar or vaginal HPV-associated lesion defined as ≥ cervical intraepithelial neoplasia grade 2(CIN2) ) , Vulvar intraepithelial neoplasia grade 2 (VIN2), vaginal intraepithelial neoplasia grade 2 (VaIN2 ) or invasive carcinoma
* Previous vaccination against HPV (at least one dose)
* Ongoing or planned pregnancy foreseen in the next 7 months
* Other immunodeficiency conditions such as ongoing or previous (within 6 months) chemotherapy against cancer or chronic systemic corticosteroids treatment or immunosuppressive therapy after transplantation
* Any condition contraindicating intramuscular injection such as warfarin therapy.

Ages: 15 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — only female will be included
Enrollment: 170 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2023-05-02 (Actual); Study Completion 2028-05-02 (Estimated)

PRIMARY OUTCOMES:
Rate of seroconversion in HPV antibodies against HPV | Month 7
  The rate of seroconversion of specific neutralizing antibodies against each HPV vaccine genotypes (6/11/16/18/31/33/45/52/58) one month after completion of a three doses schedule (0, 2 and 6 months) in women seronegative at baseline for these antibodies.

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (Safety and tolerability of the vaccines). | day 2 to 7 after each vaccine administration
  It will be evaluated by a specific questionnaire on a phone call made by the research team to the participant and scheduled at least 48 hours and maximum 7 days after each vaccine dose; the questionnaire will evaluate whether there is any complain regarding local reaction (pain, redness, swelling, pruritus), systemic reaction (fever, malaise and fatigue) or other side effect. In case of any usual complain > mild stage, or the presence of an unusual complain, the patient will be assessed by a visit and physical examination performed by the research team. The questionnaire has been elaborated according to the published data on safety evaluation of the 9-valent vaccine.
Impact of vaccine administration on T-lymphocyte CD4+ cell count and HIV viremia | Month 7
  The potential impact of vaccine administration on T-lymphocyte CD4+ cell count and HIV viremia will be assessed by measuring CD4 cell count and HIV viremia at baseline (any measure within 6 months before screening can be taken into account) and month 7. Any detectable HIVRNA >50 cp/ml will be reassessed on a second samples taken 2-4 weeks later. Any significant decrease in T-lymphocyte CD4+ cell count (defined as a decrease by more of 5% in the percentage or >100 cells/µl) will be reassessed on a second sample taken 2-4 weeks later.
Measure of the geometric mean titre of specific neutralizing antibodies against each HPV vaccine genotypes (6/11/16/18/31/33/45/52/58). | Month 7
  The measure of the geometric mean titre of specific neutralizing antibodies against each HPV vaccine genotypes (6/11/16/18/31/33/45/52/58) will be assessed before vaccination and 1 month after vaccination completion.
Cellular immune response | Month 7
  The cellular immune response will be evaluated in a subset of 40 patients (aged 18-40 years old) by measuring specific CD4+T cells expressing CD40, IL2, IFN-g or TNF-alpha against HPV 16/18/31/52 and 58. The analysis will be performed on a PMBC sample; a separate IC has to be signed for this sub-analysis
Incidence and prevalence rates of HPV infections | Month 18, 24,36,48 and 60
  Detection of HPV will be performed by molecular technique by the national reference center for HPV (AML, Antwerpen), performed on cervical swab taken by the gynecologist at baseline and month 18. The baseline gynecological sample might have been taken up to 6 months before the vaccination. These swabs will be sampled in all participants with previous vaginal sexually activity. In case of no previous vaginal sexual intercourse, the samples will not be taken.
The incidence and prevalence rates of abnormal cervical cytology | Month 18
  Cervical cytology will be performed by by the national reference center for HPV (AML, Antwerpen) on cervical swab taken by the gynecologist at baseline and month 18. The baseline gynecological sample might have been taken up to 12 months before the vaccination. These swabs will be sampled in all participants with previous vaginal sexually activity. In case of no previous vaginal sexual intercourse, the samples will not be taken.
Completion of vaccine schedule. | Month 7
  Rate of patients with completion of their vaccine schedule.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Konopnicki, MD, PhD, Principal Investigator — Centre Hospitalier Universitaire Saint Pierre
Locations (1):
- Service de Maladies Infectieuses, CHU Saint-Pierre, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Yes
Supporting Information: Study Protocol, ICF
Time Frame: within 12 months of the study completion

DOCUMENTS (2):
  • Study Protocol (2023-12-15): https://cdn.clinicaltrials.gov/large-docs/21/NCT03391921/Prot_001.pdf
  • Informed Consent Form (2020-07-22): https://cdn.clinicaltrials.gov/large-docs/21/NCT03391921/ICF_000.pdf